CLINICAL TRIAL: NCT00575081
Title: Physiological Brain Atlas Development
Acronym: Brain Atlas
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dario Englot, Assistant Professor, Neurosurgery Department, Vanderbilt University Medical Center
Other Study IDs: 060232; 1R01EB006136-01 (NIH); 2R01EB006136 (NIH); 1R41NS063705-01A1 (NIH); 9R42MH100007-03 (NIH)
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease; Obsessive Compulsive Disorder; Dystonia; Essential Tremor; Epilepsy
Keywords: Physiological Brain Atlas, Brain registry, Brain database
MeSH Terms: conditions — Parkinson Disease; Obsessive-Compulsive Disorder; Dystonia; Essential Tremor; Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stereotactic Brain Procedures: Patients who have consented to undergo or have undergone a stereotactic brain procedure for any reason including those who need Deep Brain Stimulation, SEEG or other brain neurmodulation device implant.
  Interventions: Device: Stereotactic brain procedures

INTERVENTIONS:
Device: Stereotactic brain procedures — Stereotactic brain procedures

SUMMARY:
The NIH grant has funded the development of a physiological brain atlas registry that will allow us to significantly improve the data collectioin and use of physiological data into a normalized brain volume. This initially was used to improve DBS implants for Parkinson's Disease, Dystonia, Essential Tremor, and OCD, but now includes data acquired during all stereotactic brain procedures.

DETAILED DESCRIPTION:
Purpose:

1. To create a brain atlas that will allow physiological and clinical information to be assigned to anatomical locations in MRI space, utilizing non-rigid MRI normalization algorithms. These data will specifically be acquired from the population of patients undergoing stereotactic brain procedures.
2. To collate and analyze the brain data placed in the atlas in a statistical manner that allows doctors to understand and treat brain disease more precisely and based on population data. For example, this would allow surgeons to predict optimal targeting locations for DBS implants, neurologists to program implants based on multiple physiological variables, including pre-operative severity of disease, intraoperative neurophysiological observations, and post-operative responses to previous therapies in a larger population of subjects.
3. To allow precise relationships to be visualized in one anonymized MRI volume, which can lead to new findings across larger populations of subjects in the field of brain science.
4. To locate all the data in a HIPAA compliant, anonymized location that clinicians and researchers can access securely without compromising personal healthcare information (PHI).

Protocol:

1. Patients who have consented to undergo or have undergone a stereotactic brain procedure for any reason will be asked to participate in this study.
2. Permission from the patient will be sought to allow the entry of all related data to be entered into the atlas database. Specifically, this includes any and all related pre-operative, intra-operative, and post-operative clinical, radiographic, and psychologic testing done for the purposes of the surgery.
3. The data must be entered in a confidential fashion and secured within a section of the database that can be accessed only by persons authorized to view patient healthcare information (PHI). Persons authorized to enter and view individual PHI must have taken and passed the CITI certification and presented documentation of this credential to the IRB study investigator (Dr. Konrad) or his Clinical Trials Specialist (Melba Isom).
4. Access to individual patient data within the database can be done through a secure login linked to the person's qualifications to access PHI. The list of authorized persons (such as treating physicians and members of the surgical team) will be determined by Dr. Konrad and updated at least on an annual basis within the database by Dr. Dawant. Dr. Dawant will be responsible to ensure that PHI is physically and virtually secure within the atlas database.
5. Once in the database, patient identifiers will be codified and not accessible for any queries outside of those certified in step 3. Non-patient specific information can be analyzed, sorted or queried in response to specific statistical questions by any investigator of the research team or authorized person, as designated by the database developer (Dr. Dawant) or his designee.
6. Data contained within the atlas will be analyzed and regularly reported to members of the Atlas research team regarding accurate display and representation of the data.
7. Clinical and physiological data will continue to be entered for every subject who consents to participate in this study for the duration of their care.
8. If subjects no longer wish to have their data tracked within the atlas, they can call the study coordinator (Melba Isom) and have their name removed from any further data collection from the time of notification forward. All previously collected data will still be accessible and not expunged from the database.
9. We plan to recruit 5,000 patients from Vanderbilt and participating sites.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are recommended for Stereotactic Brain procedures
* Any patient who has agreed to undergo a Stereotactic Brain procedure
* Patients age under 6 -90 years old

Exclusion Criteria:

* Patients who fail recommendation for Stereotactic Brain procedures
* Patients not consented for Stereotactic Brain procedures
* Patients outside the age range of 6 -90 years old
* Patients or legal guardians not able to provide informed consent

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have already consented to having a stereotactic brain procedure for surgical treatment or implantation of a device to treat any brain disease. This includes patients who are undergoing normal neurosurgical care for the treatment of their movement disorder (like tremor and Parkinson's disease), epilepsy, pain, or psychiatric disease.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To create an atlas that will allow physiological information to be assigned to anatomical locations in MRI space, utilizing non-rigid MRI normalization algorithms. | life of study
  The above data will specifically be acquired from the population of patients undergoing Stereotactic Brain Surgery

SECONDARY OUTCOMES:
To collate and analyze the physiological atlas in a statistical manner that allows doctors to understand and treat brain disease more precisely and based on population data. | life of study
  This is based on multiple physiological variables, including pre-operative severity of disease, intraoperative neurophysiological observations, and post-operative response to DBS stimulation therapy and brain disease requiring stereotactic procedures

OTHER OUTCOMES:
Assist surgical team intro-operatively | life of study
  Assist the surgical team intro-operatively in making adjustments in the final DBS target location based on knowledge gained from population data contained within the atlas.
Improve post-implant programming of DBS unit | life of study
  Improve post-implant programming of the DBS unit based on atlas predictions of optimal zones of therapy; to allow precise relationships to be gvisualized in one anonymized MRI volume, which can lead to new findings across larger populations of subjects in the field of brain science

CONTACTS AND LOCATIONS:
Overall Officials: Darioq j Englot, MD, Ph.D., Principal Investigator — Vanderbilt University, Dept. Neurosurgery
Locations (1):
- Vanderbilt Univeristy, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided